CLINICAL TRIAL: NCT03862352
Title: Glasgow Natural History Study Of Covered Coronary Interventions
Acronym: GNOCCI
Status: Completed | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Responsible Party: Principal Investigator, Dr Thomas J Ford, Clinical Research Fellow | Honorary Fellow (Interventional Cardiology), NHS National Waiting Times Centre Board
Other Study IDs: 1.0
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Perforation; Coronary Stent Occlusion; Stent Thrombosis
Keywords: Coronary artery perforation; Covered coronary stent; Calcific coronary disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary artery perforation (iatrogenic): Any coronary artery perforation defined according to the Ellis criteria.
  Interventions: Device: Covered coronary stent

INTERVENTIONS:
Device: Covered coronary stent — Insertion of covered coronary stent as part of standard care

SUMMARY:
Covered stents (CS) are a potentially lifesaving treatment for grade III coronary perforation but delivery can be challenging, and the long-term durability and safety including risk of acute stent thrombosis are unknown. The GNOCCI study aims to evaluate long term outcomes after coronary perforation including patients treated with covered stents.

DETAILED DESCRIPTION:
Covered stents (CS) are a potentially lifesaving treatment for grade III coronary perforation but delivery can be challenging, and the long-term durability and safety including risk of acute stent thrombosis are unknown. Using an electronic data base, details of all coronary perforations are identified and anonymised patient and procedural details are recorded.Procedural major adverse cardiac events (pMACE) are defined as a composite of death, myocardial infarction, stroke, target vessel revascularization or cardiac surgery within 24 hours of the index procedure. Two independent cardiologists adjudicate outcomes and differences in opinion are resolved by consensus with a third cardiologist.

The overall GNOCCI study aims are:

1. Evaluate procedural and long term outcomes after coronary perforation
2. Long term safety and clinical events in patients treated with covered stents.

ELIGIBILITY:
Inclusion Criteria:

* Any coronary artery perforation during percutaneous coronary intervention

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients undergoing invasive coronary angiography with planned myocardial revascularisation using percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Procedural major adverse cardiac events (pMACE) | 24 hours of the index procedure.
  Defined as a composite of death, myocardial infarction, stroke, target vessel revascularization or cardiac surgery

SECONDARY OUTCOMES:
MACE | Up to 10 years
  death, myocardial infarction, stroke, target vessel revascularization or cardiac surgery
Stent thrombosis | Up to 10 years
  ARC definite or probable
Unsuccessful covered stent deployment | 24 hours of the index procedure.
  Attempted covered stent insertion without sealing of perforation, defined by case review of two independent cardiologists from source files

CONTACTS AND LOCATIONS:
Overall Officials: Tom J Ford, MBChB (Hons), Principal Investigator — GJNH/University of Glasgow
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Contact PI for data sharing

REFERENCES:
- [Derived] Ford TJ, Adamson C, Morrow AJ, Rocchiccioli P, Collison D, McCartney PJ, Shaukat A, Lindsay M, Good R, Watkins S, Eteiba H, Robertson K, Berry C, Oldroyd KG, McEntegart M. Coronary Artery Perforations: Glasgow Natural History Study of Covered Stent Coronary Interventions (GNOCCI) Study. J Am Heart Assoc. 2022 Oct 4;11(19):e024492. doi: 10.1161/JAHA.121.024492. Epub 2022 Sep 21. PMID 36129052